CLINICAL TRIAL: NCT06832774
Title: Exploration of Treatment Effect of Novel Hormone Therapy Combined with Local Treatment Based on PSMA PET/CT Evaluation in MHSCP Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Han Bangmin, Chief physician, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025-009
Record Dates: First submitted 2025-01-19; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer Metastatic Disease
MeSH Terms: interventions — Gonadotropin-Releasing Hormone; abiraterone; apalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Novel hormone therapy (Active Comparator)
  Interventions: Drug: Gonadotropin releasing hormone analog (GnRHa) + Novel hormone therapy (abiraterone, apalutamide or rezvilutamide).
- Novel hormone therapy and Local treatment (Experimental)
  Interventions: Procedure: Local treatment; Drug: Gonadotropin releasing hormone analog (GnRHa) + Novel hormone therapy (abiraterone, apalutamide or rezvilutamide).

INTERVENTIONS:
Procedure: Local treatment — For bone lesions, radiotherapy or orthopedic surgery may be selected. For lymph node lesions, radiotherapy or high-energy focused ultrasound (HIFU) maybe selected. The specific treatment plan will be determined by the researcher and based on the patient's clinical condition.
  Arms: Novel hormone therapy and Local treatment
Drug: Gonadotropin releasing hormone analog (GnRHa) + Novel hormone therapy (abiraterone, apalutamide or rezvilutamide). — The intervention contains gonadotropin releasing hormone analog (GnRHa) and novel hormone therapy. For GnRHa, there are 3 options available. 1. "Leuprorelin"/"Prostap" or "Staladex". 2. "Goserelin"/"Zoladex". 3. "Triptorelin" /"LiverTox". For novel hormone therapy, there are also 3 options available. 1. "Abiraterone"/ "ZYTIGA®". 2. "Apalutamide"/"ERLEADA®". 3. "Rezvilutamide"/"ARIANE®". The specific treatment plan will be designed according to patients' clinical conditions based on EAU guidelines.

SUMMARY:
At present, there is still controversy over the treatment of metastatic hormone sensitive prostate cancer (mHSPC). Major guidelines and consensus suggest that novel hormone therapy (NHT) should be used as the basic treatment for mHSPC, and metastasis directed therapy can be combined depending on the clinical situation. However, it is still unclear how to develop more specific and individualized treatment plans for mHSPC patients. On the other hand, prostate-specific membrane antigen (PSMA) which is highly specifically expressed in prostate epithelial cells has been widely used as a PET/CT target for the diagnosis and staging of prostate cancer. However, there is still a lack of clinical evidence on how to use it to guide the treatment of prostate cancer. Therefore, this study intends to include patients diagnosed with mHSPC by PSMA PET/CT. After 6 months of NHT, PSMA PET/CT will be re-evaluated and patients with remaining active lesions on PSMA PET/CT will be included for randomization. The aim of this study is to explore the effect of NHT combined with local treatment on delaying disease progression and prolonging survival in patients with active lesions on PSMA PET/CT after NHT, providing new insights into the treatment of mHSCP patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients over the age of 18;
2. The physical condition (PS) score of the Eastern Cooperative Oncology Group (ECOG) is 0, 1, or 2 points;
3. Expected lifespan >2 years;
4. All newly diagnosed patients with metastatic prostate cancer (mHSPC, metastatic hormone sensitive prostate cancer) diagnosed by PSMA PET/CT, and still present active lesions on PSMA PET/CT after receiving new endocrine therapy;
5. Has not received any other treatment for prostate cancer before;
6. No significant organ dysfunction upon evaluation;
7. Agreed to sign the written consent form for this study, indicating a comprehensive understanding of the purpose and process of this study, and willingness to participate in this study.

Exclusion Criteria:

1. A medical history of any other active malignant tumor within 2 years (excluding fully treated basal cell or squamous cell skin cancer, superficial bladder cancer or any other cancer in situ that is currently in complete remission);
2. Prostate biopsy shows sarcomatoid cells, ductal carcinoma, or neuroendocrine cell components;
3. Severe complications, immune suppression, severe mental illness, severe activity restriction, or inability to comply with this study;
4. Currently participating in other clinical trials for prostate cancer;
5. According to the researcher's judgment, there are conditions that are not in line with the best interests of the subjects participating in the study, or may hinder, limit, or interfere with the study protocol.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival, PFS | From enrollment to the end of treatment at 12 weeks
  Progression includes biochemical progression, clinical progression, and imaging progression. The definition of biochemical progression is a PSA increase of more than 25% and an absolute increase of 2ng/ml compared above baseline or nadir. The definition of clinical progression is the emergence of any new clinical symptoms related to the primary and metastatic lesions of prostate cancer. The definition of imaging progression is the appearance of any new metastatic lesion in CT/MR/PET/CT scan. When one of the above criteria is met, it can be considered as disease progression.